CLINICAL TRIAL: NCT06214780
Title: Effect of Heatwaves on Glycemic Control in Adult Patients With Type 1 Diabetes Mellitus Treated With Advanced Hybrid Closed Loop Systems
Brief Title: Effect of Heatwaves on Glycemic Control in People With Type 1 Diabetes Treated With Artificial Pancreas
Acronym: HEAT1
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: CI
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: advanced hybrid closed-loop; artificial pancreas; heatwave; climate change; global warming
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Type 1 diabetes patients: Adult patients treated with advanced hybrid closed-loop in Castilla-La Mancha during summer 2023.
  Interventions: Device: advanced hybrid closed-loop

INTERVENTIONS:
Device: advanced hybrid closed-loop — An advanced hybrid closed-loop system is a type of insulin delivery system that uses an algorithm to automatically adjust insulin delivery based on glucose levels. It combines an insulin pump with a continuous glucose monitor (CGM) and uses a closed-loop algorithm to adjust insulin doses based on real-time glucose readings. The "hybrid" aspect refers to the fact that the system still requires some user input, such as entering meal information, but the algorithm takes over the majority of insulin dosing decisions.

SUMMARY:
To analyze the effect of heatwaves on interstitial glucose in adult patients with type 1 diabetes mellitus treated with artificial pancreas

DETAILED DESCRIPTION:
Observational retrospective study to analyze the effect of heatwaves on interstitial glucose in adult patients with type 1 diabetes mellitus treated with advanced hybrid closed-loop systems in the Castilla-La Mancha region (southcentral Spain). Main objective is the difference in time in range of intersticial glucose between 3.0-10 mmol/L (70-180 mg/d) measured throught real-time continuous glucose monitoring during the two consecutive greatest heatwave during summer 2024 (5th-26th August) comparted to the following period (27th August to 17th September). Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant. The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Older than 18 years old
* Using advanced hybrid closed-loop systems (AHCL)
* Paired active AHCL data from the heatwave periods and two consecutive weeks

Exclusion Criteria:

* Younger than 18 years old
* Not using AHCL
* Not having active paired AHCL data from the analyzed periods

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult type 1 diabetes patients using AHCL during and after heatwaves in Castilla-La Mancha (Spain).
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in time in range | 14 days
  Change in Time in range (TIR) 3.0-10 mmol/L (70-180 mg/d) of interstitial glucose from the heatwaves period to 14 days after its end

SECONDARY OUTCOMES:
Adherence to advaced hybrid closed-loop | 14 days
  Change in Time of use automatization of advanced hybrid closed-loop (% possible time of use) from the heatwaves period to 14 days after its end
Change in Time below range 1 (TBR1) | 14 days
  Change in Time bellow range <3.9 mmol/L (<70 mg/dL) of the interstitial glucose from the heatwaves period to 14 days after its endfrom the heatwave period to 14 days after its end
Change in Time below range 2 (TBR2) | 14 days
  Change in Time bellow range <3 mmol/L (<54 mg/dL) of the interstitial glucose from the heatwaves period to 14 days after its end
Change in Time above range 1 (TAR1) | 14 days
  Change in Time above range >10 mmol/L(>180 mg/dL) of the interstitial glucose from the heatwaves period to 14 days after its end
Change in Time above range 2 (TAR2) | 14 days
  Change in Time above range >13.9 mmol/L (>250 mg/dL) of the interstitial glucose from the heatwaves period to 14 days after its end
Change in Coefficient of variation percentage (CV) | 14 days
  Change in Coefficient of variation percentage of interstitial glucose from the heatwaves period to 14 days after its end
Change in Glucose management index | 14 days
  Change in Glucose management index of interstitial glucose from the heatwaves period to 14 days after its end
Change in Time in hypoglycemia | 14 days
  Change in Daily time in hypoglycemia (<3.9 mmol/L, <70 mg/dL) of interstitical glucose from the heatwaves period to 14 days after its end
Change in Percentage of patients attaining the the International Consensus on Time in Range (ICTR) goals | 14 days
  Change in Percentage of patients (from total) attaining TIR>70%, TBR1<4%, TBR2<1%, TAR1<25%, TAR2<5% and CV <36% from the heatwaves period to 14 days after its end
Change in Percentage of time of varibles modes of automatization | 14 days
  Change in Percentage of time of varibles modes of automatization (temporal objective, sleeping mode, exercise mode) from the heatwaves period to 14 days after its end

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - La Mancha-Centro Hospital, Alcázar de San Juan, Ciudad Real
  - Santa Barbara Hospital, Puertollano, Ciudad Real
  - Valdepeñas General Hospital, Valdepeñas, Ciudad Real
  - Virgen del Prado Hospital, Talavera de la Reina, Toledo
  - Albacete University Hospital, Albacete
  - Ciudad Real General University Hospital, Ciudad Real
  - Virgen de la Luz University Hospital, Cuenca
  - Guadalajara University Hospital, Guadalajara
  - Toledo University Hospital, Toledo

IPD SHARING:
Plan to Share IPD: No
Under other researchers request.

REFERENCES:
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Song X, Jiang L, Zhang D, Wang X, Ma Y, Hu Y, Tang J, Li X, Huang W, Meng Y, Shi A, Feng Y, Zhang Y. Impact of short-term exposure to extreme temperatures on diabetes mellitus morbidity and mortality? A systematic review and meta-analysis. Environ Sci Pollut Res Int. 2021 Nov;28(41):58035-58049. doi: 10.1007/s11356-021-14568-0. Epub 2021 Jun 8. PMID 34105073
- [Background] Moon J. The effect of the heatwave on the morbidity and mortality of diabetes patients; a meta-analysis for the era of the climate crisis. Environ Res. 2021 Apr;195:110762. doi: 10.1016/j.envres.2021.110762. Epub 2021 Jan 27. PMID 33515577
- [Background] Moreno-Fernandez J, Sastre J, Herranz S, Pines P, Gomez FJ, Quiroga I, Moya AJ, Gonzalvo C, Miralles R, Calderon-Vicente D, Palma M, Gargallo J, Munoz-Rodriguez JR. Effect of the historic Spanish heatwave over glycemic control in adult patients with type 1 diabetes. Sci Total Environ. 2023 Sep 1;889:164045. doi: 10.1016/j.scitotenv.2023.164045. Epub 2023 May 17. PMID 37201805
- See also: Spanish national forecast service — https://www.aemet.es/es/serviciosclimaticos/cambio_climat